CLINICAL TRIAL: NCT05972811
Title: Investigation of the Effect of Cold Application on Pain Caused by Jackson Pratt Drain Removal in Patients With Kidney Transplantation
Brief Title: The Effect of Cold Application on Pain Developed Due to Drain Removal in Patients With Kidney Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Ufuk Akkurt, PhD (c), Department of Nursing, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Karadeniz T. Uni.
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Pain
Keywords: Pain; Pain Management; Kidney Transplantation; Drainage; Cryotherapy
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Prospective, parallel randomized controlled clinical trial
Who Masked: Care Provider
Masking Description: The application will be made by the researcher. However, pain assessment will be done by the nurse who cares for the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold application (Experimental): A frozen ice pack at -10 °C will be prepared for the patients in the experimental group. With these ice packs, the JP will be cooled to 13.6 °C, taking into account the literature, in order to create a local anesthetic effect on the drain outlet area before the drain is removed. Skin temperature will be measured intermittently with an infrared thermometer. When the skin temperature reaches 13.6 °C, the doctor will be informed and the drain will be removed. Before starting the cold application, immediately after the drain is removed, and after 15 minutes, considering the literature, pain will be measured with the "Visual Analog Scale". By ensuring that the drain removal procedure is performed by the same physician, individual differences that may arise will be prevented.
  Interventions: Other: Cold application
- Control (No Intervention): No treatment will be applied to the patients in the control group. Pain measurement will be made with Visual Analog Scale before drain removal, immediately after drain removal, and 15 minutes later.

INTERVENTIONS:
Other: Cold application — In the experimental group, cold application will be made until the skin temperature of the drain exit area reaches 13.6 °C. And before drain removal, immediately after drain removal and 15 minutes later, pain levels will be measured with VAS and analgesic needs will be questioned
  Arms: Cold application

SUMMARY:
The study was planned as a prospective, randomized controlled study to examine the effect of cold application on pain due to Jackson Pratt drain removal in kidney transplant patients.

DETAILED DESCRIPTION:
During kidney transplant surgery, a Jackson Pratt Drain (JP) is placed in the surgical field to monitor lymphocele and urinary leakage. This drain is a closed system that opens outward from the skin at a point close to the incision line. This drain is removed by pulling when the drainage amount falls below 30 ml. This procedure is known to cause serious pain. In our study, which was planned as a prospective, randomized controlled study, it was aimed to examine the effect of cold application in the pain caused by the removal of the JP drain in patients with kidney transplantation. The population of the study will be patients who had a kidney transplant in İstinye University Hospital Liv Hospital Organ Transplant Center (n=76). In the study, patients will be assigned to the experimental and control groups by the block randomization method. "Patient Information Form" and "Visual Analog Scale" (VAS) will be used as data collection tools. In the experimental group, cold application will be made until the skin temperature of the drain exit area reaches 13.6 °C. Then, the drain removal process will be performed by the physician. In the control group, no application will be made. In both study groups before drain removal, immediately after drain removal and 15 minutes later, pain levels will be measured with VAS and analgesic needs will be questioned. Chi-square and t-tests will be used to compare demographic data in the analysis process of the data. ANOVA test will be applied to compare pain scores between groups.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* Being conscious, oriented to person, place and time,
* No history of mental pathology,
* No history of drug or alcohol use,
* Having a body mass index of <30 kg/m2,
* Not using any analgesic or sedative medication one hour before drain removal.

Exclusion Criteria:

* IV analgesic or sedative treatment during cold application,
* Having a history of chronic pain,
* Having previous drain removal experience,
* Anxiety,
* Refusal to participate in the research,
* Unstable hemodynamic status.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Pain evaluated using the Visual Analog Scale (VAS) | Pain measurement will be made with VAS just before drain removal, immediately after drain removal, and 15 minutes later.
  According to this scale, "0" indicates no pain, "1-4" indicates mild pain, "5-6" indicates moderate pain, and "7-10" indicates severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek ÇİLİNGİR, Professor, Study Director — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No